CLINICAL TRIAL: NCT06273943
Title: Impact of Long-acting Injectable Cabotegravir for HIV Pre-exposure Prophylaxis Persistence and Coverage in Men Who Have Sex With Men in France: a Randomized Controlled Clinical Trial.
Brief Title: Impact of Long-acting Injectable Cabotegravir for HIV PrEP in MSM in France.
Acronym: CABOPrEP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 0410s CABOPrEP; 2024-510678-25 (EudraCT Number)
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Prevention
Keywords: HIV pre-exposure prophylaxis; PrEP; MSM; Long-acting injectable; cabotegravir; TDF/FTC; Persistence
MeSH Terms: interventions — cabotegravir; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to remain on their current oral PrEP regimen with daily and/or on-demand TDF/FTC (Control arm) or to switch to a CAB-LA based PrEP (Intervention arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral PrEP with daily or on-demand TDF/FTC (Active Comparator): Participants randomly assigned to the oral PrEP regimen will be instructed to take a single dose combination of TDF 300 mg + FTC 200 mg (TDF/FTC), either daily or on-demand, according to their preferences.
  Interventions: Drug: Tenofovir disoproxil/Emtricitabine 300mg/200mg fixed-dose combination tablets, for oral use; Procedure: Rectal Biopsies
- Long-acting injectable PrEP with cabotegavir (Experimental): Participants assigned to the cabotegravir group will initially take a 30mg oral tablet of cabotegravir daily for a four-week period. Following this initial phase, they will receive 13 intramuscular injections of 600mg (3mL) long-acting injectable cabotegravir (CAB-LA) administered every two months after an initial loading dose given one month after the last oral tablet.
  Interventions: Drug: Cabotegravir Tablets, for oral use.; Drug: Cabotegravir Extended-Release Injectable Suspension, for intramuscular use.; Procedure: Rectal Biopsies

INTERVENTIONS:
Drug: Cabotegravir Tablets, for oral use. — Participants randomly assigned to the cabotegravir arm will be instructed to take by mouth a single tablet of cabotegavir 30mg once daily for four weeks.
  Other Names: VOCABRIA
  Arms: Long-acting injectable PrEP with cabotegavir
Drug: Cabotegravir Extended-Release Injectable Suspension, for intramuscular use. — Participants will receive 600mg (3mL) CAB LA injections intramuscularly at Month 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24. The injections will be performed in the gluteal muscle by trained healthcare providers at study sites.
  Other Names: APRETUDE
  Arms: Long-acting injectable PrEP with cabotegavir
Drug: Tenofovir disoproxil/Emtricitabine 300mg/200mg fixed-dose combination tablets, for oral use — * Daily regimen: a single tablet of TDF/FTC every 24 hours, regardless of sexual activity. If PrEP was stopped, resume with two pills of TDF/FTC followed by one pill every 24 hours.
  * On-demand regimen: a loading dose of two pills of TDF/FTC 2 to 24 hours before sexual intercourse, a third pill 24 hours after the first drug intake and a fourth pill 24 hours later. In case of daily sexual intercourse, participants will be instructed to take one pill per day until the last sexual intercourse, then to take the two post-exposure pills. If the last dose of TDF/FTC was taken less than one week prior, a leading dose with a single pill of TDF/FTC is sufficient.
  Other Names: TRUVADA
  Arms: Oral PrEP with daily or on-demand TDF/FTC
Procedure: Rectal Biopsies — This intervention concerns only participants involved in the rectal tissue HIV-1 permissibility sub-study.
  The proctologist collects ten rectal biopsies at different time points before and after PrEP initiation according to the randomization arm.

SUMMARY:
The purpose of this study is to evaluate if offering long-acting injectable cabotegravir (CAB-LA) as an additional HIV prevention choice among oral PrEP-experienced men who have sex with men (MSM) in France can significantly increase the sustained PrEP use over time and the PrEP coverage of at-risk sexual risk behaviors.

DETAILED DESCRIPTION:
Long-acting injectable cabotegravir (CAB-LA) is a promising agent to address the issue of uptake, adherence, and persistence among oral PrEP users who faced adherence challenges. However, the potential benefits of offering CAB-LA as an additional prevention option for MSM adherent to oral PrEP has yet to be demonstrated. We hypothesize that offering CAB-LA as an additional prevention option for MSM already using oral PrEP can mitigate PrEP fatigue over time, resulting in enhanced PrEP use and increased coverage of at-risk sexual intercourses.

This study is designed as a pragmatic, open-label, multicenter, parallel-group, randomized controlled clinical trial aiming to enroll MSM using PrEP for at least 6 months. Participants will be randomly assigned in a 1:1 ratio to remain on their current oral PrEP regimen with daily and/or on-demand TDF/FTC (Control arm) or to switch to a CAB-LA based PrEP (Intervention arm). Participants will be enrolled over 6 months and followed for two years. The trial will be conducted at 9 clinical sites in the Paris region. The primary objective of the study will be to compare the sustained PrEP use over time among participants randomized to CAB-LA vs. oral TDF/FTC based PrEP at Months 12 and 24. The main secondary objectives will aim to evaluate the PrEP coverage of at-risk sexual intercourses, the change from baseline in sexual risk behaviors, the safety of the drugs, and the HIV incidence.

The study protocol includes three ancillary studies:

* Social science: Focus groups will be conducted among study participants to investigate their perceptions of CAB-LA, motivations for using it, adherence and persistence, changes in HIV risk perception, and impact on sexual satisfaction. Additionally, this study will assess healthcare providers' perceptions, barriers, and facilitators regarding CAB-LA implementation for PrEP.
* Rectal tissue HIV-1 permissibility: This study aims to evaluate the protection from HIV-1 at different time points after oral and injectable CAB initiation using a model of Ex-vivo rectal tissue and PBMCs infection with HIV-1.
* Medico-economics analysis: The main objective of this study is to establish cost-effectiveness performance benchmarks for CAB-LA in HIV PrEP.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years.
* Cisgender men who have sex with men.
* Have taken oral TDF/FTC based PrEP during the past 6 months, either daily or on-demand, with a documented PrEP prescription.
* Agreeing to be contacted personally by telephone (call, SMS) or e-mail.
* Person affiliated with or a beneficiary of a social security scheme (article L1121-11 of the Public Health Code).
* Informed and written consent, signed by the person and the investigator on the day of inclusion, at the latest, and before any examination carried out within the setting of the study (article L1122-1-1 of the Public Health Code).

Non-inclusion criteria

* Positive HIV test result at screening or enrollment visit, even if HIV infection is not confirmed.
* Symptoms and/or clinical signs consistent with an acute HIV infection.
* History of seizure disorder.
* Ongoing Post-Exposure Prophylaxis (PEP) for HIV.
* Last titer of hepatitis B surface antibody (anti-HBs) < 10 mIU/mL.
* Concomitant use of antimycobacterial (rifampin, rifapentine) or enzyme-inducing anticonvulsants (carbamazepine, oxcarbazepine, phenobarbital, phenytoin, etc.).
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Participants having a non-treated chronic HCV infection.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) > 5-fold the upper normal limit (UNL).
* Creatinine clearance lower than 50mL/min.
* History of chronic renal disease, osteoporosis or osteopenia.
* Inflammatory skin conditions which compromise the safety of intramuscular (IM) injections.
* Known thrombocytopenia or any other known bleeding disorder, which would contraindicate IM injection.
* Treatment with oral anticoagulant (antiplatelet agents are allowed).
* Known or suspected allergy to study product components.
* Surgically placed buttock implants.
* Planned trip abroad of more than 2 consecutive months or planned move outside the Ile de France region.
* Individuals who, upon the investigator's judgement, will not be likely to comply the clinical trial procedures, or with any condition incompatible with study participation.
* Person participating in another research study with an exclusion period still in progress at inclusion. Participants in the ANRS PREVENIR study are authorized to participate in the ANRS CABOPrEP trial.
* Person under guardianship or curatorship or deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Men
Enrollment: 322 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of protocol visits completed with a documented PrEP prescription aligned with the randomization arm. | At Month 12

SECONDARY OUTCOMES:
Number of protocol visits completed with a documented PrEP prescription aligned with the randomization arm. | At Month 24
Number of participants with missing follow-up visits, temporary PrEP discontinuation, permanent PrEP discontinuation, switching to another PrEP regimen, study discontinuation, lost to follow-up. | At 12 and 24 Months.
Number of participants whose last condomless anal sexual intercourse was not covered by PrEP. | At each study visits.
Number of condomless anal sexual intercourse in the month prior to each study visit. | At each study visits.
Number of sexual partners in the last 3 months. | At baseline, 6, 12, 18 and 24 months
Mean PrEP satisfaction score based on study arm. | At baseline, 6, 12, 18 and 24 months.
Number of participants with syphilis, chlamydiae, and/or gonorrhea infection. | From Day 1 up to end of study.
Number of participants with Grade 2 or higher clinical or laboratory drug-related adverse events at any time during the study. | From Day 1 up to end of study.
Change from baseline in body weight (kg). | At Months 12 and 24.
Change from baseline in lipids | At Months 12 and 24.
  Fasting total Cholesterol (mmol/L), LDL cholesterol (mmol/L), HDL cholesterol (mmol/L).
Change from baseline in the insulin resistance index (HOMA-IR). | At Months 12 and 24.
  HOMA-IR : [fasting glucose (mmol/L) × fasting insulin (μmol/L)/22.5]
Number and severity of injection site reaction. | After 12 and 24 Months.
Cabotegravir concentration in plasma and tenofovir diphosphate and emtricitabine triphosphate concentration in dried blood spots. | At baseline, 6, 12, 18 and 24 months.
Number of participants with new HIV infection. | From Day 1 up to end of study.
Number of participants who used psychoactive drugs in the last 3 months | At baseline, 6, 12, 18 and 24 months.
Score of quality of life measured by the EuroQol-5D questionnaire | At baseline, 6, 12, 18 and 24 months.
  The possible range of scores is 0 to 100%, with the higher scores indicating better outcome.
Depression score assessed with the Center for Epidemiologic Studies Depression Scale (CES-D). | At baseline,12, and 24 months.
  The possible range of scores is 0 to 60, with the higher scores indicating worse outcome.
Self-esteem score assessed with the Rosenberg scale. | At baseline,12, and 24 months.
  The scale ranges from 0 to 30, with the higher score indicating a better outcome.
Number and nature of uses of community peer support and therapeutic patient education. | At baseline, 6, 12, 18 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Molina, Professor, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (8):
- France (8):
  - Hôpital Hôtel Dieu, Paris, Île-de-France Region
  - Hôpital Lariboisière, Paris, Île-de-France Region
  - Hôpital Saint Louis, Paris, Île-de-France Region
  - Hôpital Saint Antoine, Paris, Île-de-France Region
  - Hôpital La Pitié Salpêtrière, Paris, Île-de-France Region
  - Hôpital Necker, Paris, Île-de-France Region
  - Hôpital Bichat, Paris, Île-de-France Region
  - Hôpital Tenon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No